CLINICAL TRIAL: NCT04276623
Title: Identifying Atopic Dermatitis Patients at Risk for Developing Conjunctivitis During Dupilumab Treatment
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: UMC Utrecht (Other)
Collaborators: Sanofi (Industry)
Responsible Party: Principal Investigator, Dr M.S. de Bruin-Weller, Principle Investigator, UMC Utrecht
Other Study IDs: 18/537
Record Dates: First submitted 2020-02-10; First posted 2020-02-19 (Actual); Last update posted 2023-11-29 (Actual); Status verified 2023-11

CONDITIONS: Atopic Dermatitis
Keywords: Dupilumab; Dupixent; Conjunctivitis; Bioday
MeSH Terms: conditions — Dermatitis, Atopic; Conjunctivitis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Blood, tear fluid, impression cytology of the conjunctiva
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Study on ophthalmological comorbidities and the underlying pathomechanisms of conjunctivitis during dupilumab treatment in atopic dermatitis (AD) patients. Patients participate in the Bioday Registry.

ELIGIBILITY:
Inclusion Criteria:

* Adult patients with atopic dermatitis indicated for dupilumab, without current use of oral immunosuppressive treatment .

Exclusion Criteria:

* Treatment with oral or ocular immunosuppressive drugs 2 weeks prior to start of dupilumab treatment

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adult patients with atopic dermatitis indicated for dupilumab, without current use of oral immunosuppressive treatment .
Sampling Method: Probability Sample
Enrollment: 150 (Estimated)
Dates: Start 2020-02-25 (Actual); Primary Completion 2023-12-31 (Estimated); Study Completion 2023-12-31 (Estimated)

PRIMARY OUTCOMES:
Relationship between goblet cell density and the incidence of conjunctivitis over time | change of goblet cell density between baseline, 4 weeks and 28 weeks after start dupilumab, at the moment of the development of eye symptoms, 4 weeks after ocular treatment
  Establish the relationship between goblet cell densitiy and the incidence of conjunctivitis during dupilumab treatment in AD patients. Goblet cell density will determined by counting the goblet cells. The amount of goblet cells will be compared at different time points. Goblet cells will be collected using Impression Cytology of the conjunctiva and will be stained directly.
Relationship between goblet cell density and the risk of conjunctivitis | change of goblet cell density between baseline, 4 weeks and 28 weeks after start dupilumab, at the moment of the development of eye symptoms, 4 weeks after ocular treatment
  Establish the relationship between goblet cell densitiy and the risk of conjunctivitis during dupilumab treatment in AD patients. Goblet cell density will determined by counting the goblet cells. The amount of goblet cells will be compared at different time points. Goblet cells will be collected using Impression Cytology of the conjunctiva and will be stained directly.

SECONDARY OUTCOMES:
Conjunctival changes during dupilumab treatment using Impression Cytology | baseline, 4 weeks and 28 weeks after start dupilumab, at the moment of the development of eye symptoms, 4 weeks after ocular treatment
  Better understanding of conjunctival changes using Impression Cytology of the conjunctiva, collected at different time points during treatment with dupilumab in AD patients
Optimal treatment of conjunctivitis | at the moment of the development of eye symptoms, 4 weeks after ocular treatment
  Establish the most optimal treatment of conjunctivitis during dupilumab treatment. Ophthalmological examination will be compared at all time points to determine if the prescribed therapy is effective and optimal.

CONTACTS AND LOCATIONS:
Locations (1):
- University Medical Center Utrecht, Utrecht, Netherlands